CLINICAL TRIAL: NCT00530894
Title: THE PARTNER TRIAL: Placement of AoRTic TraNscathetER Valve Trial Edwards SAPIEN Transcatheter Heart Valve
Brief Title: THE PARTNER TRIAL: Placement of AoRTic TraNscathetER Valve Trial
Acronym: PARTNER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-06-US
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Critical Aortic Stenosis
Keywords: Valvular Heart Disease; Critical/Severe Aortic Stenosis; High risk symptomatic patients
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Cohort A: Sapien Valve
  Interventions: Device: Edwards SAPIEN Transcatheter Heart Valve
- 2 (Active Comparator): Cohort A: other surgical valve
  Interventions: Device: Surgical Valve Replacement
- 3 (Experimental): Cohort B: Sapien Valve
  Interventions: Device: Edwards SAPIEN Transcatheter Heart Valve
- 4 (Active Comparator): Cohort B: Medical therapy
  Interventions: Other: medical management and/or balloon aortic valvuloplasty

INTERVENTIONS:
Device: Edwards SAPIEN Transcatheter Heart Valve
  Arms: 1; 3
Device: Surgical Valve Replacement
  Arms: 2
Other: medical management and/or balloon aortic valvuloplasty
  Arms: 4

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the device and delivery systems (transfemoral and transapical) in high risk, symptomatic patients with severe aortic stenosis.

DETAILED DESCRIPTION:
Subjects will undergo a physical exam and screening tests will be performed to determine if they are either A) a patient with a high surgical risk or B) not a candidate for surgery. They will then be randomized (like the flip of a coin) to have the investigational device implanted or to receive the current surgical or medical management available.

ELIGIBILITY:
Inclusion Criteria Cohort A

1. Patients must have co-morbidities such that the surgeon and cardiologist Co-PIs concur that the predicted risk of operative mortality is ≥15% and/or a minimum STS score of 10
2. Patient has senile degenerative aortic valve stenosis with echocardiographically derived criteria: mean gradient >40 mmHg or jet velocity greater than 4.0 m/s or an initial aortic valve area of < 0.8 cm2
3. Patient is symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA Functional Class II or greater
4. The subject or the subject's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the IRB of the respective clinical site
5. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits

   Cohort B All candidates for Cohort B of this study must meet #2, 3, 4, 5 of the above criteria and
6. The subject, after formal consults by a cardiologist and two cardiovascular surgeons agree that medical factors preclude operation, based on a conclusion that the probability of death or serious, irreversible morbidity exceeds the probability of meaningful improvement. Specifically, the probability of death or serious, irreversible morbidity should exceed 50%.

Exclusion Criteria

1. Evidence of an acute myocardial infarction ≤ 1month before the intended treatment.
2. Aortic valve is a congenital unicuspid or bicuspid valve; or is non-calcified
3. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+).
4. Any therapeutic invasive cardiac procedure performed within 30 days of the index procedure, (or 6 months if the procedure was a drug eluting coronary stent implantation).
5. Pre-existing prosthetic heart valve in any position, prosthetic ring, or severe (greater than 3+) mitral insufficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1057 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Principal Investigator — New York-Presbyterian Hospital/Columbia University Medical Center; Craig Smith, MD, Principal Investigator — New York-Presbyterian Hospital/Columbia University Medical Center
Locations (26):
- United States (22):
  - Scripps Memorial Hospital/Scripps Green Hospital, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Ochsner Clinic, New Orleans, Louisiana
  - Boston Mass General, Boston, Massachusetts
  - Brigham and Women's, Boston, Massachusetts
  - Mayo Clinic-Saint Marys Hospital, Rochester, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Barnes-Jewish/Washington University, St Louis, Missouri
  - New York Presbyterian Hospital - Cornell, New York, New York
  - Columbia University Medical Center, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical City Dallas, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
- Canada (3):
  - Vancouver St. Paul's, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Laval Hospital, Québec
- Heart Center Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Huded CP, Arnold SV, Chhatriwalla AK, Saxon JT, Kapadia S, Yu X, Webb JG, Thourani VH, Kodali SK, Smith CR, Mack MJ, Leon MB, Cohen DJ. Rehospitalization Events After Aortic Valve Replacement: Insights From the PARTNER Trial. Circ Cardiovasc Interv. 2022 Dec;15(12):e012195. doi: 10.1161/CIRCINTERVENTIONS.122.012195. Epub 2022 Dec 20. PMID 36538580
- [Derived] Shahim B, Redfors B, Lindman BR, Chen S, Dahlen T, Nazif T, Kapadia S, Gertz ZM, Crowley AC, Li D, Thourani VH, Kodali SK, Zajarias A, Babaliaros VC, Guyton RA, Elmariah S, Herrmann HC, Cohen DJ, Mack MJ, Smith CR, Leon MB, George I. Neutrophil-to-Lymphocyte Ratios in Patients Undergoing Aortic Valve Replacement: The PARTNER Trials and Registries. J Am Heart Assoc. 2022 Jun 7;11(11):e024091. doi: 10.1161/JAHA.121.024091. Epub 2022 Jun 3. PMID 35656983
- [Derived] Vincent F, Thourani VH, Ternacle J, Redfors B, Cohen DJ, Hahn RT, Li D, Crowley A, Webb JG, Mack MJ, Kapadia S, Russo M, Smith CR, Alu MC, Leon MB, Pibarot P. Time-of-Day and Clinical Outcomes After Surgical or Transcatheter Aortic Valve Replacement: Insights From the PARTNER Trials. Circ Cardiovasc Qual Outcomes. 2022 Jan;15(1):e007948. doi: 10.1161/CIRCOUTCOMES.121.007948. Epub 2022 Jan 18. PMID 35041482
- [Derived] Summers MR, Leon MB, Smith CR, Kodali SK, Thourani VH, Herrmann HC, Makkar RR, Pibarot P, Webb JG, Leipsic J, Alu MC, Crowley A, Hahn RT, Kapadia SR, Tuzcu EM, Svensson L, Cremer PC, Jaber WA. Prosthetic Valve Endocarditis After TAVR and SAVR: Insights From the PARTNER Trials. Circulation. 2019 Dec 10;140(24):1984-1994. doi: 10.1161/CIRCULATIONAHA.119.041399. Epub 2019 Nov 6. PMID 31690104
- [Derived] Kapadia SR, Huded CP, Kodali SK, Svensson LG, Tuzcu EM, Baron SJ, Cohen DJ, Miller DC, Thourani VH, Herrmann HC, Mack MJ, Szerlip M, Makkar RR, Webb JG, Smith CR, Rajeswaran J, Blackstone EH, Leon MB; PARTNER Trial Investigators. Stroke After Surgical Versus Transfemoral Transcatheter Aortic Valve Replacement in the PARTNER Trial. J Am Coll Cardiol. 2018 Nov 13;72(20):2415-2426. doi: 10.1016/j.jacc.2018.08.2172. PMID 30442284
- [Derived] Elmariah S, Fearon WF, Inglessis I, Vlahakes GJ, Lindman BR, Alu MC, Crowley A, Kodali S, Leon MB, Svensson L, Pibarot P, Hahn RT, Thourani VH, Palacios IF, Miller DC, Douglas PS, Passeri JJ; PARTNER Trial Investigators and PARTNER Publications Office. Transapical Transcatheter Aortic Valve Replacement Is Associated With Increased Cardiac Mortality in Patients With Left Ventricular Dysfunction: Insights From the PARTNER I Trial. JACC Cardiovasc Interv. 2017 Dec 11;10(23):2414-2422. doi: 10.1016/j.jcin.2017.09.023. PMID 29217004
- [Derived] Douglas PS, Leon MB, Mack MJ, Svensson LG, Webb JG, Hahn RT, Pibarot P, Weissman NJ, Miller DC, Kapadia S, Herrmann HC, Kodali SK, Makkar RR, Thourani VH, Lerakis S, Lowry AM, Rajeswaran J, Finn MT, Alu MC, Smith CR, Blackstone EH; PARTNER Trial Investigators. Longitudinal Hemodynamics of Transcatheter and Surgical Aortic Valves in the PARTNER Trial. JAMA Cardiol. 2017 Nov 1;2(11):1197-1206. doi: 10.1001/jamacardio.2017.3306. PMID 28973520
- [Derived] Lindman BR, Otto CM, Douglas PS, Hahn RT, Elmariah S, Weissman NJ, Stewart WJ, Ayele GM, Zhang F, Zajarias A, Maniar HS, Jilaihawi H, Blackstone E, Chinnakondepalli KM, Tuzcu EM, Leon MB, Pibarot P. Blood Pressure and Arterial Load After Transcatheter Aortic Valve Replacement for Aortic Stenosis. Circ Cardiovasc Imaging. 2017 Jul;10(7):e006308. doi: 10.1161/CIRCIMAGING.116.006308. PMID 28701528
- [Derived] Beohar N, Doshi D, Thourani V, Jensen H, Kodali S, Zhang F, Zhang Y, Davidson C, McCarthy P, Mack M, Kapadia S, Leon M, Kirtane A. Association of Transcatheter Aortic Valve Replacement With 30-Day Renal Function and 1-Year Outcomes Among Patients Presenting With Compromised Baseline Renal Function: Experience From the PARTNER 1 Trial and Registry. JAMA Cardiol. 2017 Jul 1;2(7):742-749. doi: 10.1001/jamacardio.2017.1220. PMID 28467527
- [Derived] Daubert MA, Weissman NJ, Hahn RT, Pibarot P, Parvataneni R, Mack MJ, Svensson LG, Gopal D, Kapadia S, Siegel RJ, Kodali SK, Szeto WY, Makkar R, Leon MB, Douglas PS. Long-Term Valve Performance of TAVR and SAVR: A Report From the PARTNER I Trial. JACC Cardiovasc Imaging. 2016 Dec 8:S1936-878X(16)30895-6. doi: 10.1016/j.jcmg.2016.11.004. Online ahead of print. PMID 28017714
- [Derived] Kapadia S, Agarwal S, Miller DC, Webb JG, Mack M, Ellis S, Herrmann HC, Pichard AD, Tuzcu EM, Svensson LG, Smith CR, Rajeswaran J, Ehrlinger J, Kodali S, Makkar R, Thourani VH, Blackstone EH, Leon MB. Insights Into Timing, Risk Factors, and Outcomes of Stroke and Transient Ischemic Attack After Transcatheter Aortic Valve Replacement in the PARTNER Trial (Placement of Aortic Transcatheter Valves). Circ Cardiovasc Interv. 2016 Sep;9(9):e002981. doi: 10.1161/CIRCINTERVENTIONS.115.002981. PMID 27601428
- [Derived] Anjan VY, Herrmann HC, Pibarot P, Stewart WJ, Kapadia S, Tuzcu EM, Babaliaros V, Thourani VH, Szeto WY, Bavaria JE, Kodali S, Hahn RT, Williams M, Miller DC, Douglas PS, Leon MB. Evaluation of Flow After Transcatheter Aortic Valve Replacement in Patients With Low-Flow Aortic Stenosis: A Secondary Analysis of the PARTNER Randomized Clinical Trial. JAMA Cardiol. 2016 Aug 1;1(5):584-92. doi: 10.1001/jamacardio.2016.0759. PMID 27437665
- [Derived] Suri RM, Minha S, Alli O, Waksman R, Rihal CS, Satler LP, Greason KL, Torguson R, Pichard AD, Mack M, Svensson LG, Rajeswaran J, Lowry AM, Ehrlinger J, Mick SL, Tuzcu EM, Thourani VH, Makkar R, Holmes D, Leon MB, Blackstone EH. Learning curves for transapical transcatheter aortic valve replacement in the PARTNER-I trial: Technical performance, success, and safety. J Thorac Cardiovasc Surg. 2016 Sep;152(3):773-780.e14. doi: 10.1016/j.jtcvs.2016.04.028. Epub 2016 Apr 13. PMID 27215927
- [Derived] Kodali S, Williams MR, Doshi D, Hahn RT, Humphries KH, Nkomo VT, Cohen DJ, Douglas PS, Mack M, Xu K, Svensson L, Thourani VH, Tuzcu EM, Weissman NJ, Leon M, Kirtane AJ. Sex-Specific Differences at Presentation and Outcomes Among Patients Undergoing Transcatheter Aortic Valve Replacement: A Cohort Study. Ann Intern Med. 2016 Mar 15;164(6):377-84. doi: 10.7326/M15-0121. Epub 2016 Feb 23. PMID 26903039
- [Derived] Beohar N, Kirtane AJ, Blackstone E, Waksman R, Holmes D Jr, Minha S, Alli O, Suri RM, Svensson LG, Leon M, Kodali S. Trends in Complications and Outcomes of Patients Undergoing Transfemoral Transcatheter Aortic Valve Replacement: Experience From the PARTNER Continued Access Registry. JACC Cardiovasc Interv. 2016 Feb 22;9(4):355-363. doi: 10.1016/j.jcin.2015.10.050. Epub 2016 Jan 20. PMID 26803420
- [Derived] Biviano AB, Nazif T, Dizon J, Garan H, Fleitman J, Hassan D, Kapadia S, Babaliaros V, Xu K, Parvataneni R, Rodes-Cabau J, Szeto WY, Fearon WF, Dvir D, Dewey T, Williams M, Mack MJ, Webb JG, Miller DC, Smith CR, Leon MB, Kodali S. Atrial Fibrillation Is Associated With Increased Mortality in Patients Undergoing Transcatheter Aortic Valve Replacement: Insights From the Placement of Aortic Transcatheter Valve (PARTNER) Trial. Circ Cardiovasc Interv. 2016 Jan;9(1):e002766. doi: 10.1161/CIRCINTERVENTIONS.115.002766. PMID 26733582
- [Derived] Lindman BR, Zajarias A, Maniar HS, Miller DC, Suri RM, Arnold SV, Webb J, Svensson LG, Kodali S, Xu K, Ayele GM, Lin F, Wong SC, Babaliaros V, Thourani VH, Douglas PS, Lim S, Leon MB, Mack MJ. Risk stratification in patients with pulmonary hypertension undergoing transcatheter aortic valve replacement. Heart. 2015 Oct;101(20):1656-64. doi: 10.1136/heartjnl-2015-308001. Epub 2015 Aug 11. PMID 26264371
- [Derived] Dizon JM, Nazif TM, Hess PL, Biviano A, Garan H, Douglas PS, Kapadia S, Babaliaros V, Herrmann HC, Szeto WY, Jilaihawi H, Fearon WF, Tuzcu EM, Pichard AD, Makkar R, Williams M, Hahn RT, Xu K, Smith CR, Leon MB, Kodali SK; PARTNER Publications Office. Chronic pacing and adverse outcomes after transcatheter aortic valve implantation. Heart. 2015 Oct;101(20):1665-71. doi: 10.1136/heartjnl-2015-307666. Epub 2015 Aug 10. PMID 26261157
- [Derived] Thourani VH, Jensen HA, Babaliaros V, Kodali SK, Rajeswaran J, Ehrlinger J, Blackstone EH, Suri RM, Don CW, Aldea G, Williams MR, Makkar R, Svensson LG, McCabe JM, Dean LS, Kapadia S, Cohen DJ, Pichard AD, Szeto WY, Herrmann HC, Devireddy C, Leshnower BG, Ailawadi G, Maniar HS, Hahn RT, Leon MB, Mack M. Outcomes in Nonagenarians Undergoing Transcatheter Aortic Valve Replacement in the PARTNER-I Trial. Ann Thorac Surg. 2015 Sep;100(3):785-92; discussion 793. doi: 10.1016/j.athoracsur.2015.05.021. Epub 2015 Aug 1. PMID 26242213
- [Derived] Szeto WY, Svensson LG, Rajeswaran J, Ehrlinger J, Suri RM, Smith CR, Mack M, Miller DC, McCarthy PM, Bavaria JE, Cohn LH, Corso PJ, Guyton RA, Thourani VH, Lytle BW, Williams MR, Webb JG, Kapadia S, Tuzcu EM, Cohen DJ, Schaff HV, Leon MB, Blackstone EH; Placement of Aortic Transcatheter Valves Trial Investigators. Appropriate patient selection or health care rationing? Lessons from surgical aortic valve replacement in the Placement of Aortic Transcatheter Valves I trial. J Thorac Cardiovasc Surg. 2015 Sep;150(3):557-68.e11. doi: 10.1016/j.jtcvs.2015.05.073. Epub 2015 Jun 30. PMID 26238287
- [Derived] Gada H, Kirtane AJ, Wang K, Lei Y, Magnuson E, Reynolds MR, Williams MR, Kodali S, Vahl TP, Arnold SV, Leon MB, Thourani V, Szeto WY, Cohen DJ; PARTNER Investigators. Temporal Trends in Quality of Life Outcomes After Transapical Transcatheter Aortic Valve Replacement: A Placement of AoRTic TraNscathetER Valve (PARTNER) Trial Substudy. Circ Cardiovasc Qual Outcomes. 2015 Jul;8(4):338-46. doi: 10.1161/CIRCOUTCOMES.114.001335. Epub 2015 Jun 9. PMID 26058718
- [Derived] Green P, Arnold SV, Cohen DJ, Kirtane AJ, Kodali SK, Brown DL, Rihal CS, Xu K, Lei Y, Hawkey MC, Kim RJ, Alu MC, Leon MB, Mack MJ. Relation of frailty to outcomes after transcatheter aortic valve replacement (from the PARTNER trial). Am J Cardiol. 2015 Jul 15;116(2):264-9. doi: 10.1016/j.amjcard.2015.03.061. Epub 2015 Apr 18. PMID 25963221
- [Derived] Blackstone EH, Suri RM, Rajeswaran J, Babaliaros V, Douglas PS, Fearon WF, Miller DC, Hahn RT, Kapadia S, Kirtane AJ, Kodali SK, Mack M, Szeto WY, Thourani VH, Tuzcu EM, Williams MR, Akin JJ, Leon MB, Svensson LG. Propensity-matched comparisons of clinical outcomes after transapical or transfemoral transcatheter aortic valve replacement: a placement of aortic transcatheter valves (PARTNER)-I trial substudy. Circulation. 2015 Jun 2;131(22):1989-2000. doi: 10.1161/CIRCULATIONAHA.114.012525. Epub 2015 Apr 1. PMID 25832034
- [Derived] Mack MJ, Leon MB, Smith CR, Miller DC, Moses JW, Tuzcu EM, Webb JG, Douglas PS, Anderson WN, Blackstone EH, Kodali SK, Makkar RR, Fontana GP, Kapadia S, Bavaria J, Hahn RT, Thourani VH, Babaliaros V, Pichard A, Herrmann HC, Brown DL, Williams M, Akin J, Davidson MJ, Svensson LG; PARTNER 1 trial investigators. 5-year outcomes of transcatheter aortic valve replacement or surgical aortic valve replacement for high surgical risk patients with aortic stenosis (PARTNER 1): a randomised controlled trial. Lancet. 2015 Jun 20;385(9986):2477-84. doi: 10.1016/S0140-6736(15)60308-7. Epub 2015 Mar 15. PMID 25788234
- [Derived] Kapadia SR, Leon MB, Makkar RR, Tuzcu EM, Svensson LG, Kodali S, Webb JG, Mack MJ, Douglas PS, Thourani VH, Babaliaros VC, Herrmann HC, Szeto WY, Pichard AD, Williams MR, Fontana GP, Miller DC, Anderson WN, Akin JJ, Davidson MJ, Smith CR; PARTNER trial investigators. 5-year outcomes of transcatheter aortic valve replacement compared with standard treatment for patients with inoperable aortic stenosis (PARTNER 1): a randomised controlled trial. Lancet. 2015 Jun 20;385(9986):2485-91. doi: 10.1016/S0140-6736(15)60290-2. Epub 2015 Mar 15. PMID 25788231
- [Derived] Kapadia S, Stewart WJ, Anderson WN, Babaliaros V, Feldman T, Cohen DJ, Douglas PS, Makkar RR, Svensson LG, Webb JG, Wong SC, Brown DL, Miller DC, Moses JW, Smith CR, Leon MB, Tuzcu EM. Outcomes of inoperable symptomatic aortic stenosis patients not undergoing aortic valve replacement: insight into the impact of balloon aortic valvuloplasty from the PARTNER trial (Placement of AoRtic TraNscathetER Valve trial). JACC Cardiovasc Interv. 2015 Feb;8(2):324-333. doi: 10.1016/j.jcin.2014.08.015. PMID 25700756
- [Derived] Nazif TM, Dizon JM, Hahn RT, Xu K, Babaliaros V, Douglas PS, El-Chami MF, Herrmann HC, Mack M, Makkar RR, Miller DC, Pichard A, Tuzcu EM, Szeto WY, Webb JG, Moses JW, Smith CR, Williams MR, Leon MB, Kodali SK; PARTNER Publications Office. Predictors and clinical outcomes of permanent pacemaker implantation after transcatheter aortic valve replacement: the PARTNER (Placement of AoRtic TraNscathetER Valves) trial and registry. JACC Cardiovasc Interv. 2015 Jan;8(1 Pt A):60-9. doi: 10.1016/j.jcin.2014.07.022. PMID 25616819
- [Derived] Passeri JJ, Elmariah S, Xu K, Inglessis I, Baker JN, Alu M, Kodali S, Leon MB, Svensson LG, Pibarot P, Fearon WF, Kirtane AJ, Vlahakes GJ, Palacios IF, Douglas PS; PARTNER Investigators. Transcatheter aortic valve replacement and standard therapy in inoperable patients with aortic stenosis and low EF. Heart. 2015 Mar;101(6):463-71. doi: 10.1136/heartjnl-2014-306737. Epub 2015 Jan 13. PMID 25586156
- [Derived] Genereux P, Cohen DJ, Mack M, Rodes-Cabau J, Yadav M, Xu K, Parvataneni R, Hahn R, Kodali SK, Webb JG, Leon MB. Incidence, predictors, and prognostic impact of late bleeding complications after transcatheter aortic valve replacement. J Am Coll Cardiol. 2014 Dec 23;64(24):2605-2615. doi: 10.1016/j.jacc.2014.08.052. PMID 25524339
- [Derived] Fearon WF, Kodali S, Doshi D, Fischbein MP, Yeung AC, Tuzcu EM, Rihal CS, Babaliaros V, Zajarias A, Herrmann HC, Brown DL, Mack M, Teirstein PS, Whisenant BK, Makkar R, Kapadia S, Leon MB; PARTNER Trial Investigators. Outcomes after transfemoral transcatheter aortic valve replacement: a comparison of the randomized PARTNER (Placement of AoRTic TraNscathetER Valves) trial with the NRCA (Nonrandomized Continued Access) registry. JACC Cardiovasc Interv. 2014 Nov;7(11):1245-51. doi: 10.1016/j.jcin.2014.05.033. Epub 2014 Nov 17. PMID 25459036
- [Derived] Douglas PS, Hahn RT, Pibarot P, Weissman NJ, Stewart WJ, Xu K, Wang Z, Lerakis S, Siegel R, Thompson C, Gopal D, Keane MG, Svensson LG, Tuzcu EM, Smith CR, Leon MB. Hemodynamic outcomes of transcatheter aortic valve replacement and medical management in severe, inoperable aortic stenosis: a longitudinal echocardiographic study of cohort B of the PARTNER trial. J Am Soc Echocardiogr. 2015 Feb;28(2):210-7.e1-9. doi: 10.1016/j.echo.2014.10.009. Epub 2014 Nov 20. PMID 25455544
- [Derived] Arnold SV, Lei Y, Reynolds MR, Magnuson EA, Suri RM, Tuzcu EM, Petersen JL 2nd, Douglas PS, Svensson LG, Gada H, Thourani VH, Kodali SK, Mack MJ, Leon MB, Cohen DJ; PARTNER Investigators. Costs of periprocedural complications in patients treated with transcatheter aortic valve replacement: results from the Placement of Aortic Transcatheter Valve trial. Circ Cardiovasc Interv. 2014 Dec;7(6):829-36. doi: 10.1161/CIRCINTERVENTIONS.114.001395. Epub 2014 Oct 21. PMID 25336467
- [Derived] Rodes-Cabau J, Pibarot P, Suri RM, Kodali S, Thourani VH, Szeto WY, Svensson LG, Dumont E, Xu K, Hahn RT, Leon MB. Impact of aortic annulus size on valve hemodynamics and clinical outcomes after transcatheter and surgical aortic valve replacement: insights from the PARTNER Trial. Circ Cardiovasc Interv. 2014 Oct;7(5):701-11. doi: 10.1161/CIRCINTERVENTIONS.114.001681. Epub 2014 Sep 30. PMID 25270901
- [Derived] Pibarot P, Weissman NJ, Stewart WJ, Hahn RT, Lindman BR, McAndrew T, Kodali SK, Mack MJ, Thourani VH, Miller DC, Svensson LG, Herrmann HC, Smith CR, Rodes-Cabau J, Webb J, Lim S, Xu K, Hueter I, Douglas PS, Leon MB. Incidence and sequelae of prosthesis-patient mismatch in transcatheter versus surgical valve replacement in high-risk patients with severe aortic stenosis: a PARTNER trial cohort--a analysis. J Am Coll Cardiol. 2014 Sep 30;64(13):1323-34. doi: 10.1016/j.jacc.2014.06.1195. PMID 25257633
- [Derived] Kapadia SR, Tuzcu EM, Makkar RR, Svensson LG, Agarwal S, Kodali S, Fontana GP, Webb JG, Mack M, Thourani VH, Babaliaros VC, Herrmann HC, Szeto W, Pichard AD, Williams MR, Anderson WN, Akin JJ, Miller DC, Smith CR, Leon MB. Long-term outcomes of inoperable patients with aortic stenosis randomly assigned to transcatheter aortic valve replacement or standard therapy. Circulation. 2014 Oct 21;130(17):1483-92. doi: 10.1161/CIRCULATIONAHA.114.009834. Epub 2014 Sep 9. PMID 25205802
- [Derived] Svensson LG, Blackstone EH, Rajeswaran J, Brozzi N, Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Tuzcu EM, Webb JG, Kapadia S, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Thourani VH, Pichard AD, Bavaria JE, Herrmann HC, Williams MR, Babaliaros V, Genereux P, Akin JJ; PARTNER Trial Investigators. Comprehensive analysis of mortality among patients undergoing TAVR: results of the PARTNER trial. J Am Coll Cardiol. 2014 Jul 15;64(2):158-68. doi: 10.1016/j.jacc.2013.08.1666. PMID 25011720
- [Derived] Arnold SV, Reynolds MR, Lei Y, Magnuson EA, Kirtane AJ, Kodali SK, Zajarias A, Thourani VH, Green P, Rodes-Cabau J, Beohar N, Mack MJ, Leon MB, Cohen DJ; PARTNER Investigators. Predictors of poor outcomes after transcatheter aortic valve replacement: results from the PARTNER (Placement of Aortic Transcatheter Valve) trial. Circulation. 2014 Jun 24;129(25):2682-90. doi: 10.1161/CIRCULATIONAHA.113.007477. Epub 2014 May 23. PMID 24958751
- [Derived] Beohar N, Whisenant B, Kirtane AJ, Leon MB, Tuzcu EM, Makkar R, Svensson LG, Miller DC, Smith CR, Pichard AD, Herrmann HC, Thourani VH, Szeto WY, Lim S, Fischbein M, Fearon WF, O'Neill W, Xu K, Dewey T, Mack M. The relative performance characteristics of the logistic European System for Cardiac Operative Risk Evaluation score and the Society of Thoracic Surgeons score in the Placement of Aortic Transcatheter Valves trial. J Thorac Cardiovasc Surg. 2014 Dec;148(6):2830-7.e1. doi: 10.1016/j.jtcvs.2014.04.006. Epub 2014 Apr 13. PMID 24820191
- [Derived] Williams M, Kodali SK, Hahn RT, Humphries KH, Nkomo VT, Cohen DJ, Douglas PS, Mack M, McAndrew TC, Svensson L, Thourani VH, Tuzcu EM, Weissman NJ, Kirtane AJ, Leon MB. Sex-related differences in outcomes after transcatheter or surgical aortic valve replacement in patients with severe aortic stenosis: Insights from the PARTNER Trial (Placement of Aortic Transcatheter Valve). J Am Coll Cardiol. 2014 Apr 22;63(15):1522-8. doi: 10.1016/j.jacc.2014.01.036. Epub 2014 Feb 19. PMID 24561149
- [Derived] Genereux P, Cohen DJ, Williams MR, Mack M, Kodali SK, Svensson LG, Kirtane AJ, Xu K, McAndrew TC, Makkar R, Smith CR, Leon MB. Bleeding complications after surgical aortic valve replacement compared with transcatheter aortic valve replacement: insights from the PARTNER I Trial (Placement of Aortic Transcatheter Valve). J Am Coll Cardiol. 2014 Mar 25;63(11):1100-9. doi: 10.1016/j.jacc.2013.10.058. Epub 2013 Nov 27. PMID 24291283
- [Derived] Lindman BR, Pibarot P, Arnold SV, Suri RM, McAndrew TC, Maniar HS, Zajarias A, Kodali S, Kirtane AJ, Thourani VH, Tuzcu EM, Svensson LG, Waksman R, Smith CR, Leon MB. Transcatheter versus surgical aortic valve replacement in patients with diabetes and severe aortic stenosis at high risk for surgery: an analysis of the PARTNER Trial (Placement of Aortic Transcatheter Valve). J Am Coll Cardiol. 2014 Mar 25;63(11):1090-9. doi: 10.1016/j.jacc.2013.10.057. Epub 2013 Nov 27. PMID 24291272
- [Derived] Elmariah S, Palacios IF, McAndrew T, Hueter I, Inglessis I, Baker JN, Kodali S, Leon MB, Svensson L, Pibarot P, Douglas PS, Fearon WF, Kirtane AJ, Maniar HS, Passeri JJ; PARTNER Investigators. Outcomes of transcatheter and surgical aortic valve replacement in high-risk patients with aortic stenosis and left ventricular dysfunction: results from the Placement of Aortic Transcatheter Valves (PARTNER) trial (cohort A). Circ Cardiovasc Interv. 2013 Dec;6(6):604-14. doi: 10.1161/CIRCINTERVENTIONS.113.000650. Epub 2013 Nov 12. PMID 24221391
- [Derived] Makkar RR, Jilaihawi H, Mack M, Chakravarty T, Cohen DJ, Cheng W, Fontana GP, Bavaria JE, Thourani VH, Herrmann HC, Pichard A, Kapadia S, Babaliaros V, Whisenant BK, Kodali SK, Williams M, Trento A, Smith CR, Teirstein PS, Cohen MG, Xu K, Tuzcu EM, Webb JG, Leon MB. Stratification of outcomes after transcatheter aortic valve replacement according to surgical inoperability for technical versus clinical reasons. J Am Coll Cardiol. 2014 Mar 11;63(9):901-11. doi: 10.1016/j.jacc.2013.08.1641. Epub 2013 Oct 23. PMID 24161334
- [Derived] Barbanti M, Webb JG, Hahn RT, Feldman T, Boone RH, Smith CR, Kodali S, Zajarias A, Thompson CR, Green P, Babaliaros V, Makkar RR, Szeto WY, Douglas PS, McAndrew T, Hueter I, Miller DC, Leon MB; Placement of Aortic Transcatheter Valve Trial Investigators. Impact of preoperative moderate/severe mitral regurgitation on 2-year outcome after transcatheter and surgical aortic valve replacement: insight from the Placement of Aortic Transcatheter Valve (PARTNER) Trial Cohort A. Circulation. 2013 Dec 24;128(25):2776-84. doi: 10.1161/CIRCULATIONAHA.113.003885. Epub 2013 Oct 23. PMID 24152861
- [Derived] Dvir D, Waksman R, Barbash IM, Kodali SK, Svensson LG, Tuzcu EM, Xu K, Minha S, Alu MC, Szeto WY, Thourani VH, Makkar R, Kapadia S, Satler LF, Webb JG, Leon MB, Pichard AD. Outcomes of patients with chronic lung disease and severe aortic stenosis treated with transcatheter versus surgical aortic valve replacement or standard therapy: insights from the PARTNER trial (placement of AoRTic TraNscathetER Valve). J Am Coll Cardiol. 2014 Jan 28;63(3):269-79. doi: 10.1016/j.jacc.2013.09.024. Epub 2013 Oct 16. PMID 24140659
- [Derived] Green P, Cohen DJ, Genereux P, McAndrew T, Arnold SV, Alu M, Beohar N, Rihal CS, Mack MJ, Kapadia S, Dvir D, Maurer MS, Williams MR, Kodali S, Leon MB, Kirtane AJ. Relation between six-minute walk test performance and outcomes after transcatheter aortic valve implantation (from the PARTNER trial). Am J Cardiol. 2013 Sep 1;112(5):700-6. doi: 10.1016/j.amjcard.2013.04.046. Epub 2013 May 29. PMID 23725996
- [Derived] Makkar RR, Jilaihawi H, Chakravarty T, Fontana GP, Kapadia S, Babaliaros V, Cheng W, Thourani VH, Bavaria J, Svensson L, Kodali S, Shiota T, Siegel R, Tuzcu EM, Xu K, Hahn RT, Herrmann HC, Reisman M, Whisenant B, Lim S, Beohar N, Mack M, Teirstein P, Rihal C, Douglas PS, Blackstone E, Pichard A, Webb JG, Leon MB. Determinants and outcomes of acute transcatheter valve-in-valve therapy or embolization: a study of multiple valve implants in the U.S. PARTNER trial (Placement of AoRTic TraNscathetER Valve Trial Edwards SAPIEN Transcatheter Heart Valve). J Am Coll Cardiol. 2013 Jul 30;62(5):418-30. doi: 10.1016/j.jacc.2013.04.037. Epub 2013 May 15. PMID 23684680
- [Derived] Herrmann HC, Pibarot P, Hueter I, Gertz ZM, Stewart WJ, Kapadia S, Tuzcu EM, Babaliaros V, Thourani V, Szeto WY, Bavaria JE, Kodali S, Hahn RT, Williams M, Miller DC, Douglas PS, Leon MB. Predictors of mortality and outcomes of therapy in low-flow severe aortic stenosis: a Placement of Aortic Transcatheter Valves (PARTNER) trial analysis. Circulation. 2013 Jun 11;127(23):2316-26. doi: 10.1161/CIRCULATIONAHA.112.001290. Epub 2013 May 9. PMID 23661722
- [Derived] Hahn RT, Pibarot P, Stewart WJ, Weissman NJ, Gopalakrishnan D, Keane MG, Anwaruddin S, Wang Z, Bilsker M, Lindman BR, Herrmann HC, Kodali SK, Makkar R, Thourani VH, Svensson LG, Akin JJ, Anderson WN, Leon MB, Douglas PS. Comparison of transcatheter and surgical aortic valve replacement in severe aortic stenosis: a longitudinal study of echocardiography parameters in cohort A of the PARTNER trial (placement of aortic transcatheter valves). J Am Coll Cardiol. 2013 Jun 25;61(25):2514-21. doi: 10.1016/j.jacc.2013.02.087. Epub 2013 Apr 23. PMID 23623915
- [Derived] Reynolds MR, Magnuson EA, Lei Y, Wang K, Vilain K, Li H, Walczak J, Pinto DS, Thourani VH, Svensson LG, Mack MJ, Miller DC, Satler LE, Bavaria J, Smith CR, Leon MB, Cohen DJ; PARTNER Investigators. Cost-effectiveness of transcatheter aortic valve replacement compared with surgical aortic valve replacement in high-risk patients with severe aortic stenosis: results of the PARTNER (Placement of Aortic Transcatheter Valves) trial (Cohort A). J Am Coll Cardiol. 2012 Dec 25;60(25):2683-92. doi: 10.1016/j.jacc.2012.09.018. Epub 2012 Nov 1. PMID 23122802
- [Derived] Green P, Woglom AE, Genereux P, Daneault B, Paradis JM, Schnell S, Hawkey M, Maurer MS, Kirtane AJ, Kodali S, Moses JW, Leon MB, Smith CR, Williams M. The impact of frailty status on survival after transcatheter aortic valve replacement in older adults with severe aortic stenosis: a single-center experience. JACC Cardiovasc Interv. 2012 Sep;5(9):974-81. doi: 10.1016/j.jcin.2012.06.011. PMID 22995885
- [Derived] Reynolds MR, Magnuson EA, Wang K, Thourani VH, Williams M, Zajarias A, Rihal CS, Brown DL, Smith CR, Leon MB, Cohen DJ; PARTNER Trial Investigators. Health-related quality of life after transcatheter or surgical aortic valve replacement in high-risk patients with severe aortic stenosis: results from the PARTNER (Placement of AoRTic TraNscathetER Valve) Trial (Cohort A). J Am Coll Cardiol. 2012 Aug 7;60(6):548-58. doi: 10.1016/j.jacc.2012.03.075. Epub 2012 Jul 18. PMID 22818074
- [Derived] Kodali SK, Williams MR, Smith CR, Svensson LG, Webb JG, Makkar RR, Fontana GP, Dewey TM, Thourani VH, Pichard AD, Fischbein M, Szeto WY, Lim S, Greason KL, Teirstein PS, Malaisrie SC, Douglas PS, Hahn RT, Whisenant B, Zajarias A, Wang D, Akin JJ, Anderson WN, Leon MB; PARTNER Trial Investigators. Two-year outcomes after transcatheter or surgical aortic-valve replacement. N Engl J Med. 2012 May 3;366(18):1686-95. doi: 10.1056/NEJMoa1200384. Epub 2012 Mar 26. PMID 22443479
- [Derived] Makkar RR, Fontana GP, Jilaihawi H, Kapadia S, Pichard AD, Douglas PS, Thourani VH, Babaliaros VC, Webb JG, Herrmann HC, Bavaria JE, Kodali S, Brown DL, Bowers B, Dewey TM, Svensson LG, Tuzcu M, Moses JW, Williams MR, Siegel RJ, Akin JJ, Anderson WN, Pocock S, Smith CR, Leon MB; PARTNER Trial Investigators. Transcatheter aortic-valve replacement for inoperable severe aortic stenosis. N Engl J Med. 2012 May 3;366(18):1696-704. doi: 10.1056/NEJMoa1202277. Epub 2012 Mar 26. PMID 22443478
- [Derived] Miller DC, Blackstone EH, Mack MJ, Svensson LG, Kodali SK, Kapadia S, Rajeswaran J, Anderson WN, Moses JW, Tuzcu EM, Webb JG, Leon MB, Smith CR; PARTNER Trial Investigators and Patients; PARTNER Stroke Substudy Writing Group and Executive Committee. Transcatheter (TAVR) versus surgical (AVR) aortic valve replacement: occurrence, hazard, risk factors, and consequences of neurologic events in the PARTNER trial. J Thorac Cardiovasc Surg. 2012 Apr;143(4):832-843.e13. doi: 10.1016/j.jtcvs.2012.01.055. PMID 22424519
- [Derived] Reynolds MR, Magnuson EA, Wang K, Lei Y, Vilain K, Walczak J, Kodali SK, Lasala JM, O'Neill WW, Davidson CJ, Smith CR, Leon MB, Cohen DJ; PARTNER Investigators. Cost-effectiveness of transcatheter aortic valve replacement compared with standard care among inoperable patients with severe aortic stenosis: results from the placement of aortic transcatheter valves (PARTNER) trial (Cohort B). Circulation. 2012 Mar 6;125(9):1102-9. doi: 10.1161/CIRCULATIONAHA.111.054072. Epub 2012 Feb 3. PMID 22308299
- [Derived] Reynolds MR, Magnuson EA, Lei Y, Leon MB, Smith CR, Svensson LG, Webb JG, Babaliaros VC, Bowers BS, Fearon WF, Herrmann HC, Kapadia S, Kodali SK, Makkar RR, Pichard AD, Cohen DJ; Placement of Aortic Transcatheter Valves (PARTNER) Investigators. Health-related quality of life after transcatheter aortic valve replacement in inoperable patients with severe aortic stenosis. Circulation. 2011 Nov 1;124(18):1964-72. doi: 10.1161/CIRCULATIONAHA.111.040022. Epub 2011 Oct 3. PMID 21969017
- [Derived] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Derived] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243

RESULTS

PARTICIPANT FLOW:
Groups:
- High Risk: TAVR; Inoperable: TAVR: Edwards SAPIEN Transcatheter Heart Valve
- High Risk: SAVR: Surgical Aortic Valve Replacement
- Inoperable: Medical Therapy: Medical management and/or balloon aortic valvuloplasty
Period: Overall Study
Arm/Group | High Risk: TAVR | High Risk: SAVR | Inoperable: TAVR | Inoperable: Medical Therapy
Started | 348 | 351 | 179 | 179
Completed | 260 | 236 | 124 | 85
Not Completed | 88 | 115 | 55 | 94
Not completed — Death | 84 | 89 | 55 | 89
Not completed — Lost to Follow-up | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 23 | 0 | 5
Not completed — Alive and censored prior to 1 year | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The inoperable and high risk groups were not randomized against each other and were essentially two separate trials, therefore the pooled mean and standard deviations do not provide meaningful data and were not reported.
Groups:
- High Risk: SAVR: Surgical Valve Replacement
- Inoperable TAVR: Edwards SAPIEN Transcatheter Heart Valve
- Total: Total of all reporting groups
Arm/Group | High Risk: TAVR | High Risk: SAVR | Inoperable TAVR | Inoperable: Medical Therapy | Total
Number analyzed (Participants) | 348 | 349 | 179 | 179 | 1055
Age, Continuous [Mean (Standard Deviation); unit: Years]
  High Risk | 83.61 (6.83) | 84.52 (6.37) | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 84.11 (6.61)
  Inoperable | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 83.12 (8.60) | 83.18 (8.29) | 83.18 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 151 | 97 | 95 | 490
  Male | 201 | 198 | 82 | 84 | 565
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2 | 0 | 5 | 0 | 7
  Black/African American | 11 | 8 | 4 | 9 | 32
  White | 324 | 328 | 165 | 162 | 979
  Hispanic | 9 | 9 | 5 | 8 | 31
  Other | 2 | 4 | 0 | 0 | 6
NYHA Class [Number; unit: Participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
  Participants
    High Risk Class II | 20 | 21 | NA — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 41
    Operable Class II | NA — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 14 | 11 | 25
    High Risk Class III or IV | 328 | 328 | NA — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 656
    Inoperable Class III or IV | NA — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 165 | 168 | 333
Quality of Life [Mean (Standard Deviation); unit: Score] — The QOL questionnaire consisted of: Kansas City Cardiomyopathy (KCCQ), EuroQOL, SF-12. The QOL questionnaire consisted of: Kansas City Cardiomyopathy (KCCQ), The Medical Outcomes Study Short-Form 12 (SF-12) - physical and metal states. KCCQ scores are on a range of 0-100, in which 100 reflects the best health status and 0 reflects the worst health status. SF-12 questionnaire was used in which 100 reflects the best health status and 0 reflects the worst health status.
  Score
    High Risk KCCQ Overall | 39.6 (21.8) | 44.5 (21.8) | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 41.88 (21.93)
    Inoperable KCCQ Overall | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 36.19 (20.52) | 34.44 (20.14) | 35.35 (20.32)
    High Risk SF-12 Physical | 29.6 (7.6) | 30.9 (8.2) | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 30.2 (7.9)
    Inoperable SF-12 Physical | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 28.23 (7.73) | 27.70 (6.89) | 28.0 (7.23)
    High Risk SF-12 Mental | 46.9 (11.5) | 47.6 (10.7) | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 47.2 (11.1)
    Inoperable SF-12 Mental | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 44.45 (12.16) | 45.23 (11.03) | 44.84 (11.5)
STS Score [Mean (Standard Deviation); unit: Percentage] — The Society of Thoracic Surgeons (STS) score measures patient risk at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  Percentage
    High Risk | 11.8 (3.3) | 11.7 (3.5) | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 11.75 (3.40)
    Inoperable | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | NA (NA) — The inoperable and high risk groups were not randomized against each other and were essentially two separate trials | 11.2 (5.8) | 11.9 (4.8) | 11.51 (5.34)

OUTCOME MEASURES:

1. Primary Outcome: Death
Description: Death from any cause.
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | High Risk: TAVR | High Risk: SAVR | Inoperable: TAVR | Inoperable: Medical Therapy
Number analyzed (Participants) | 348 | 351 | 179 | 179
participants | 84 | 89 | 55 | 89

2. Primary Outcome: Composite of Death and Recurrence Hospitalization.
Description: Death from any cause or repeat hospitalization after intervention.
Time Frame: duration of study
Population: Composite of Death and recurrence hospitalization was not a primary outcome for the High Risk groups.
Measure: Number; unit: participants
Arm/Group | Inoperable: TAVR | Inoperable: Medical Therapy
Number analyzed (Participants) | 179 | 179
participants | 76 | 126

3. Secondary Outcome: Functional Change of NYHA
Description: NYHA classification change from baseline to 1 year visit. NYHA provides a way of classifying the extent of heart failure. New York Heart Association (NYHA) is a functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest (I) as no limitations and the highest (IV) unable to carry on any physical activity without discomfort.
Time Frame: Baseline to 1 year
Population: Note that the number of participants analyzed is different from that in the participant flow as there was some missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on scale
Arm/Group | High Risk: TAVR | High Risk: SAVR | Inoperable: TAVR | Inoperable: Medical Therapy
Number analyzed (Participants) | 334 | 314 | 172 | 167
Units on scale | 2.50 [2.35 to 2.65] | 2.60 [2.45 to 2.76] | 2.88 [2.70 to 3.07] | 3.92 [3.73 to 4.11]

4. Secondary Outcome: Number of Participants With Major Adverse Cardiac and Cerebro-vascular Events (MACCE)
Description: Number of participants with MACCE definition includes death, myocardial infarction (MI), stroke and renal failure
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | High Risk: TAVR | High Risk: SAVR | Inoperable: TAVR | Inoperable: Medical Therapy
Number analyzed (Participants) | 348 | 351 | 179 | 179
participants | 93 | 97 | 61 | 93

5. Secondary Outcome: Total Hospital Days From the Index Procedure
Description: Total hospital days from the index procedure or randomization into control arm to one year post procedure or randomization.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | High Risk: TAVR | High Risk: SAVR | Inoperable: TAVR | Inoperable: Medical Therapy
Number analyzed (Participants) | 348 | 351 | 179 | 179
Days | 17.42 (19.05) | 20.14 (23.85) | 25.24 (21.11) | 17.04 (33.46)

6. Secondary Outcome: Change in Quality of Life (QOL) From Baseline to 1 Year
Description: The QOL questionnaire consisted of: Kansas City Cardiomyopathy (KCCQ), The Medical Outcomes Study Short-Form 12 (SF-12) - physical and metal states.
  KCCQ scores are on a range of 0-100, in which 100 reflects the best health status and 0 reflects the worst health status.
  SF-12 questionnaire was used in which 100 reflects the best health status and 0 reflects the worst health status.
Time Frame: Baseline and 1 Year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | High Risk: TAVR | High Risk: SAVR | Inoperable: TAVR | Inoperable: Medical Therapy
Number analyzed (Participants) | 348 | 351 | 179 | 179
Units on a scale
  KCCQ Overall | 70.0 (22.4) | 71.1 (23.0) | 69.41 (25.37) | 46.98 (24.59)
  SF-12 Physical | 36.3 (11.0) | 36.9 (10.4) | 34.85 (11.13) | 29.68 (6.47)
  SF-12 Mental | 52.0 (10.1) | 52.9 (9.7) | 53.31 (10.00) | 46.59 (11.68)

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | High Risk: TAVR | High Risk: SAVR | Inoperable: TAVR | Inoperable: Medical Therapy
Serious Adverse Events (participants affected / at risk) | 228/348 | 238/351 | 134/179 | 151/179
Other Adverse Events (participants affected / at risk) | 230/348 | 217/351 | 140/179 | 103/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk: TAVR (N=348) | High Risk: SAVR (N=351) | Inoperable: TAVR (N=179) | Inoperable: Medical Therapy (N=179)
Other (General disorders) | 91 (127) | 86 (129) | 60 (98) | 68 (105)
Infection (including Endocarditis) (Infections and infestations) | 70 (96) | 59 (74) | 35 (53) | 30 (38)
CHF (Cardiac disorders) | 50 (73) | 51 (64) | 24 (32) | 78 (102)
Respiratory Event (Respiratory, thoracic and mediastinal disorders) | 46 (66) | 61 (76) | 25 (28) | 21 (23)
Bleeding event (Vascular disorders) | 32 (33) | 38 (42) | 23 (26) | 13 (14)
Neurological event (including TIA stroke and psychomotor deficit) (Nervous system disorders) | 33 (33) | 24 (28) | 24 (28) | 7 (8)
Arrhythmia (Cardiac disorders) | 32 (34) | 38 (44) | 22 (24) | 24 (32)
Gastro-Intestinal Event (Gastrointestinal disorders) | 22 (24) | 16 (18) | 9 (9) | 7 (10)
Hemorrhagic/Vascular event (Vascular disorders) | 21 (22) | 20 (20) | 23 (24) | 9 (9)
Renal failure (Renal and urinary disorders) | 20 (21) | 26 (29) | 11 (12) | 12 (12)
Abnormal Lab Values (Investigations) | 16 (19) | 15 (17) | 12 (17) | 11 (17)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 14 (15) | 3 (3) | 5 (7)
Hypotension (Vascular disorders) | 11 (11) | 14 (14) | 9 (9) | 4 (4)
Conduction defects (Cardiac disorders) | 11 (11) | 12 (12) | 5 (5) | 4 (4)
Renal insufficiency (Renal and urinary disorders) | 8 (8) | 8 (8) | 2 (2) | 3 (3)
Angina (Vascular disorders) | 7 (9) | 4 (5) | 2 (4) | 4 (5)
Device embolization (General disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 6 (6) | 5 (5) | 3 (4) | 6 (8)
Aortic insufficiency without paravalvular leak (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 4 (4) | 0 (0) | 2 (3) | 1 (1)
Ischemia (Vascular disorders) | 4 (4) | 2 (2) | 2 (2) | 2 (2)
MI (Vascular disorders) | 4 (4) | 4 (4) | 5 (5) | 6 (6)
Hematoma (Vascular disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
Perforation or damage to myocardium (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Thromboembolism (Vascular disorders) | 4 (4) | 3 (4) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Device migration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perivalvular leak (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Valve stenosis (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) | 33 (42)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Mitral insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Access site nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk: TAVR (N=348) | High Risk: SAVR (N=351) | Inoperable: TAVR (N=179) | Inoperable: Medical Therapy (N=179)
Other (General disorders) | 133 (242) | 124 (219) | 87 (204) | 44 (80)
Abnormal Lab Values (Investigations) | 84 (128) | 84 (136) | 51 (86) | 28 (46)
Infection (including Endocarditis) (Infections and infestations) | 60 (80) | 58 (69) | 44 (57) | 34 (52)
Arrhythmia (Cardiac disorders) | 43 (49) | 78 (88) | 26 (30) | 16 (18)
Respiratory Event (Respiratory, thoracic and mediastinal disorders) | 33 (38) | 32 (35) | 15 (18) | 10 (12)
Bleeding event (Vascular disorders) | 25 (27) | 22 (25) | 16 (21) | 7 (7)
Hemorrhagic/Vascular event (Vascular disorders) | 25 (26) | 7 (7) | 20 (25) | 3 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 47 (52) | 15 (17) | 7 (7)
Gastro-Intestinal Event (Gastrointestinal disorders) | 22 (29) | 21 (22) | 13 (18) | 7 (9)
CHF (Cardiac disorders) | 18 (18) | 7 (7) | 8 (8) | 15 (17)
Hypotension (Vascular disorders) | 19 (19) | 16 (17) | 19 (22) | 8 (9)
Hematoma (Vascular disorders) | 18 (18) | 2 (2) | 24 (28) | 8 (8)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 12 (12) | 1 (1)
Valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 11 (11)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 10 (10) | 3 (3)
Neurological event (including TIA stroke and psychomotor deficit) (Nervous system disorders) | 0 (0) | 0 (0) | 10 (11) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site cannot publish or present on overall study results not yet published. PI may publish his own clinical study data subject to EW review prior submission or presentation, but data analyses of site-specific results can occur only in intervals as specified in the CSA.

Publication of site-specific results cannot include claims of device safety and effectiveness and requires EW review.